CLINICAL TRIAL: NCT05876507
Title: The Effects of Progressive Exercises on the Vital Signs and Fatigue in Patients With Renal Transplant
Brief Title: Effect of Progressive Exercise on Renal Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Seyda Uzun Yagız, Registered nurse, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA22/239
Record Dates: First submitted 2023-03-09; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Renal Transplant; Fatigue; Vital Signs; Progressive Relaxation Exercise; Nursing
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Intervention Model Description: This is a single blind, randomized controlled study. The intervention group will receive an audio record explaining progressive relaxation exercise. Then participants will undergo training about the exercises. After training, the intervention group will perform the exercises at home by their own. The exercises will be performed everyday for 4 weeks about 25-30 minutes. Principal investigator will check the participants weekly about implementation of exercises.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): Participants will receive a training about progressive relaxation exercises on the first day, then given an audio-record containing instructions about exercises. They will perform exercises at home for 4 week and revisited by the principal investigator at the 2nd and 4th week.
  Interventions: Behavioral: Progressive relaxation exercise
- Control (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Behavioral: Progressive relaxation exercise — Progressive relaxation exercises will take 25-30 minutes of patients daily.
  Arms: exercise

SUMMARY:
The goal of this interventional study is to determine the effect of progressive relaxation exercises on the vital signs and fatigue levels of patients with renal transplantation.

DETAILED DESCRIPTION:
Renal transplant patients experience intense level of fatigue as well as vital sign problems due to treatment protocol. This research is designed to determine the effect of progressive relaxation exercises on vital signs and fatigue level of patients with renal transplantation.

In this study, the participants will be randomized in a single blind manner (participant) to either intervention (4 week exercise program) or control (routine care) groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent renal transplant within one year from the beginning of the study
* Patients having no communication problems
* Patients having a smart phone either own or o family member

Exclusion Criteria:

* Patients having musculoskeletal, cardiopulmonary, or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | Change fron baseline at 4th week
  Maintaining or normalizing systolic and blood pressure within normal range (systolic: 90-140 mmHg; diastolic 60-90 mmHg)
fatigue level | Change from baseline at 4th week
  Fatigue Severity Scale is a valid and 7-point Likert type scale. Possible scores range from 9-63. Higher scores indicate high level of fatigue. A score of 36 points or over indicates severe fatigue (Change= Lower score from the scale at the end of intervention compared to baseline).
Heart rate | Change from baseline at 4th week
  Maintaining or normalizing heart rate within normal range (60 to 100 bpm)
Respiratory rate | Change from baseline at 4th week
  Maintaining or normalizing respiratory rate within normal range (12-20 breath per minute)
Body temperature | Change from baseline at 4th week
  Maintaining or normalizing body temperature within normal range (36-37 C° in tympanic measurement)
Oxygen saturation | Change from baseline at 4th week
  Maintaining or normalizing oxygen saturation within normal range (between 95%-100% by pulse oximetry)

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available. The researchers will decide later.